CLINICAL TRIAL: NCT04532320
Title: Incidence of BRUE Among the Hospitalized Infants: Towards a Change in Medical Practices?
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Noémie BERLENGI, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2020PI133
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Brief Resolved Unexplained Events (BRUE)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The malaise of the infant represents a polymorphic pathology in its clinical presentation.

Due to the young age of the patients concerned and the parental anxiety generated, hospital management is necessary, for clinical and paraclinical evaluation and monitoring.

The practice of complementary examinations is guided by personal and family history, and the precise description of the discomfort as well as clinical examination of the child and assessment of his vital parameters.

However, in view of the particular terrain represented by infants under one year of age, a number of tests are carried out systematically, and therefore empirically, because they are not guided by the clinic.

These various tests can be invasive, anxiety-provoking for parents and generate a significant additional cost during hospital management.

An evaluation of the indication and interest of these tests is necessary in order to propose a homogeneous clinical and paraclinical management of the discomfort of the infant, in particular of discomforts of type BRUE (Brief Resolved Unexplained Events), as described in the 2016 American Academy of Pediatrics (AAP) recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Infant less than one year old
* Admitted to the paediatric emergencies of the CHRU of Nancy between 11/01/2019 and 04/30/2020 for discomfort

Exclusion Criteria:

* Child over one year old
* Reasons for consultation in paediatric emergencies other than "malaise";

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infant less than one year old, admitted to the paediatric emergencies of the CHRU of Nancy between 11/01/2019 and 04/30/2020 for discomfort
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Measurement of the proportion of BRUE-type discomfort among infants hospitalized for discomfort between 11/01/2019 and 04/30/2020 | From 11/01/2019 to 04/30/2020

SECONDARY OUTCOMES:
- Assessment of the number of additional tests performed, their nature and the results found - Assessment of the child's orientation following consultation in paediatric emergencies (return home / hospitalization) - Epidemiological analysis | From 11/01/2019 au 04/30/2020

CONTACTS AND LOCATIONS:
Overall Officials: Myriam MANGIN, Interne, Study Chair — CHRU Nancy
Locations (1):
- CHRU Nancy, Hôpital d'Enfants, Nancy, Lorraine, France

REFERENCES:
- See also: Brief Resolved Unexplained Events (Formerly Apparent Life-Threatening Events) and Evaluation of Lower-Risk Infants — http://pubmed.ncbi.nlm.nih.gov/27244835/